CLINICAL TRIAL: NCT01190566
Title: PET-MR Fusion Imaging and Surrogate Marker for Prediction and Monitoring of Response to Neoadjuvant Chemotherapy in Breast Cancer Patients
Brief Title: PET-MR for Prediction and Monitoring of Response to Neoadjuvant Chemotherapy in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, Woo Kyung Moon, Professor, Seoul National University Hospital
Other Study IDs: PET-MR Breast Cancer
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Results first posted 2015-07-07 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
Keywords: Magnetic Resonance Imaging, Functional; Tomography, Positron-Emission; chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Core biopsy specimens of breast cancer
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is:

To validate the efficacy of multiparametric MRI, FDG-PET, RGD-PET, and PET-MR fusion imaging in the prediction and monitoring response to neoadjuvant chemotherapy of locally advanced breast cancer patients.

To identify the optimal combination parameters of MR spectroscopy, diffusion-weighted MRI, dynamic contrast-enhanced MRI, FDG-PET, and RGD-PET in the prediction and monitoring response to neoadjuvant chemotherapy of locally advanced breast cancer patients.

To compare the performances of dynamic contrast-enhanced MRI using parametric response map analysis versus those of pharmacokinetic parameters (Ktrans, kep, or Ve) in the early prediction of pathological responsiveness to neoadjuvant chemotherapy in breast cancer patients

DETAILED DESCRIPTION:
Enrolled women with breast cancers who had received an anthracycline-taxane regimen and subsequent surgery were prospectively enrolled. DCE-MRI and FDG-PET scan were performed before and after the 1st cycle of chemotherapy. MR imaging parameters and SUV on PET scan within a tumor were analyzed. Clinicopathologic (age, clinical tumor stage, hormonal receptor status, and surgery type) and imaging parameters were compared according to the pathological response.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed breast cancer
* Clinical stage IIb, IIIa, IIIb, IIIc
* Must have measurable disease
* Performance status of ECOG 0-2
* Adequate, bone marrow, liver, heart, and renal function
* Who did not receive chemotherapy for breast cancer
* Must agree with and signed informed consent

Exclusion Criteria:

* Prior history of cancer besides breast cancer
* Active bacterial infection
* Pregnant or lactating women
* Psychological disease or seizure
* History of arrhythmia, congestive heart failure, myocardial infarct, or unstable angina
* Male breast cancer
* Who had a pacemaker or history of open heart surgery

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients who are candidates for neoadjuvant chemotherapy, pre-treatment MRI and PET scan, post-treatment MRI and PET scan for evaluation of chemotherapy response monitoring and residual disease
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Woo Kyung Moon, M.D., Ph.D., Principal Investigator — Department of Radiology, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Cho N, Im SA, Park IA, Lee KH, Li M, Han W, Noh DY, Moon WK. Breast cancer: early prediction of response to neoadjuvant chemotherapy using parametric response maps for MR imaging. Radiology. 2014 Aug;272(2):385-96. doi: 10.1148/radiol.14131332. Epub 2014 Apr 13. PMID 24738612
- See also: Homepage of Seoul National University Hospital Biomedical Research Institute — http://bri.snuh.org/pub/_/singlecont/view.do

RESULTS

PARTICIPANT FLOW:
Groups:
- Pathologic Complete Responders (pCR): The absence of invasive tumor cells (ductal carcinoma in situ may have been present) after surgery.
- Non-pCR: The presence of invasive tumor cells (ductal carcinoma in situ may have been present) after surgery.
Period: Overall Study
Arm/Group | Pathologic Complete Responders (pCR) | Non-pCR
Started | 6 | 42
Completed | 6 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pathologic Complete Responders (pCR) | Non-pCR | Total
Number analyzed (Participants) | 6 | 42 | 48
Age, Customized [Number; unit: participants]
  40 years old or less | 2 | 9 | 11
  more than 40 years old | 4 | 33 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 42 | 48
  Male | 0 | 0 | 0
Clinical stage (American Joint Committee on Cancer 7th edition) [Number; unit: participants]
  Stage II | 2 | 8 | 10
  Stage III | 4 | 34 | 38
Estrogen receptor [Number; unit: participants]
  Negative | 5 | 16 | 21
  Positive | 1 | 26 | 27
Progesterone receptor [Number; unit: participants]
  Negative | 5 | 31 | 36
  Positive | 1 | 11 | 12
HER2 [Number; unit: participants]
  Negative | 5 | 32 | 37
  Positive | 1 | 10 | 11
Ki-67 (Cellular marker for proliferation) [Number; unit: participants]
  14% or less (low proliferation) | 2 | 28 | 30
  more than 14% (high proliferation) | 4 | 14 | 18
Immunohistochemical subtype [Number; unit: participants]
  Hormone receptor positive | 1 | 26 | 27
  Triple negative | 4 | 10 | 14
  HER2-positive | 1 | 6 | 7

OUTCOME MEASURES:

1. Primary Outcome: Patholocial Response to Chemotherapy
Description: Pathological complete response (pCR) or non-pCR
Time Frame: Post-operation
Measure: Number; unit: participants
Groups:
- Pathologic Response to Chemotherapy: Degree of pathologic response to the neoadjuvant chemotherapy
Arm/Group | Pathologic Response to Chemotherapy
Number analyzed (Participants) | 48
participants
  Pathologic completer Responders (pCR) | 6
  Non-pCR | 42

2. Secondary Outcome: Tumor Size
Description: Maximal tumor diameter measured on magnetic resonance imaging
Time Frame: baseline, completion of 1st cycle of chemotherapy
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Pathologic Complete Responders (pCR): the absence of invasive tumor cells after surgery
- Non-pCR: the presence of invasive tumor cells after surgery
Arm/Group | Pathologic Complete Responders (pCR) | Non-pCR
Number analyzed (Participants) | 6 | 42
cm
  Baseline tumor size | 4.9 (1.8) | 5.0 (2.0)
  Post-1st chemotherapy tumor size | 4.2 (1.8) | 4.5 (1.8)

3. Secondary Outcome: Tumor Volume
Description: Tumor volume measured on 3-dimensional magnetic resonance imaging
Time Frame: Baseline, post-1st chemotherapy
Measure: Mean (Standard Deviation); unit: cm3
Arm/Group | Pathologic Complete Responders (pCR) | Non-pCR
Number analyzed (Participants) | 6 | 42
cm3
  Baseline | 22.0 (18.7) | 38.9 (89.8)
  Post-1st chemotherapy | 11.0 (13.2) | 26.4 (44.4)

4. Secondary Outcome: Proportions of Voxels Within a Tumor With Increased or Decreased Signal Intensity (Parametric Response Map Signal Intensity; PRMSI)
Description: Parametric response map analysis using a software calculates the interval change of signal intensity based on a voxel-to-voxel comparison between measurements at baseline and after the first cycle of chemotherapy. PRMSI+ indicates proportions of voxels within a tumor with increased signal intensity. PRMSI- indicates proportions of voxels within a tumor with decreased signal intensity. PRMSI0 indicates proportions of voxels within a tumor with unchanged signal intensity.
Time Frame: Baseline, post-1st chemotherapy
Measure: Mean (Standard Deviation); unit: % of voxels
Arm/Group | Pathologic Complete Responders (pCR) | Non-pCR
Number analyzed (Participants) | 6 | 42
% of voxels
  PRMSI+ | 14.0 (6.5) | 40.7 (27.2)
  PRMSI- | 83.4 (7.6) | 56.4 (27.8)
  PRMSI0 | 2.7 (1.4) | 2.9 (1.5)

5. Secondary Outcome: Constant for the Transfer of the Contrast Agent From the Plasma Compartment Into the Extracellular Extravascular Space (Ktrans)
Time Frame: Baseline, post-1st chemotherapy
Measure: Mean (Standard Deviation); unit: min-1
Arm/Group | Pathologic Complete Responders (pCR) | Non-pCR
Number analyzed (Participants) | 6 | 42
min-1
  Baseline Ktrans | 0.263 (0.044) | 0.254 (0.080)
  Post-1st chemotherapy Ktrans | 0.224 (0.076) | 0.234 (0.068)

6. Secondary Outcome: Rate Constant of the Escape of the Contrast Agent From the Extracellular Extravascular Space Into the Plasma Compartment (Kep)
Time Frame: Baseline, post-1st chemotherapy
Measure: Mean (Standard Deviation); unit: min-1
Arm/Group | Pathologic Complete Responders (pCR) | Non-pCR
Number analyzed (Participants) | 6 | 42
min-1
  Baseline | 0.616 (0.262) | 0.787 (0.729)
  Post-1st chemotherapy | 0.992 (0.917) | 0.616 (0.298)

7. Secondary Outcome: Extracellular Extravascular Space Per Unit Volume of Tissue (Ve)
Time Frame: Baseline, post-1st chemotherapy
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Pathologic Complete Responders (pCR) | Non-pCR
Number analyzed (Participants) | 6 | 42
unitless
  Baseline | 0.563 (0.129) | 0.550 (0.146)
  Post-1st chemotherapy | 0.467 (0.151) | 0.557 (0.136)

8. Secondary Outcome: Total Choline Amount of the Tumor Measured on Single Voxel 1H-magnetic Resonance Spectroscopy
Description: Single voxel 1H-magnetic resonance spectroscopy quantifies the amount of total choline-containing compounds of a tumor, which indicates cellular proliferation and malignant transformation.
Time Frame: Baseline, post-1st chemotherapy
Population: Of the 48 participants, 13 participants did not undergo magnetic resonance spectroscopy examinations due to workflow problem. We included the available data from 35 participants.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Pathologic Complete Responders (pCR) | Non-pCR
Number analyzed (Participants) | 6 | 29
unitless
  Baseline | 15.0 (8.4) | 13.5 (11.5)
  Post-1st chemotherapy | 3.4 (2.8) | 7.8 (6.3)

9. Secondary Outcome: Standardized Uptake Value on 18F-fluoro-deoxy-glucose Positron Emission Tomography
Time Frame: Baseline, post-1st chemotherapy
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Pathologic Complete Responders (pCR) | Non-pCR
Number analyzed (Participants) | 6 | 29
unitless
  Baseline | 18.9 (12.1) | 10.7 (5.6)
  Post-1st chemotherapy | 9.7 (10.7) | 7.6 (4.4)

ADVERSE EVENTS:
Time Frame: Baseline, post-1st chemotherapy, preoperative timing
Arm/Group | Pathologic Complete Responders (pCR) | Non-pCR
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/42
Other Adverse Events (participants affected / at risk) | 0/6 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No